CLINICAL TRIAL: NCT04524039
Title: Intermittent Theta Burst Stimulation (iTBS) for the Treatment of Depression in Patients With Multiple Sclerosis: a Randomized Controlled Study
Brief Title: iTBS Study for Depression in Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wei Qiu, Professor, MD, Ph.D, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-113-01
Record Dates: First submitted 2020-08-02; First posted 2020-08-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Multiple Sclerosis; Depression, Anxiety
Keywords: Multiple Sclerosis; Depression; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Multiple Sclerosis; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iTBS stimulation (Experimental): iTBS stimulation to left dorsolateral prefrontal cortex (DLPFC), twice daily, 10 days
  Interventions: Device: intermittent theta burst stimulation using a MagPro X100
- sham iTBS stimulation (Sham Comparator): sham iTBS stimulation to left dorsolateral prefrontal cortex (DLPFC), twice daily, 10 days
  Interventions: Device: sham intermittent theta burst stimulation using a MagPro X100

INTERVENTIONS:
Device: intermittent theta burst stimulation using a MagPro X100 — Patients randomized to receive iTBS in left dorsolateral prefrontal cortex, each treatment will consist of 600 stimuli (triplet 50 Hz bursts, repeated at 5 Hz; 2 s on and 8 s off; total duration of 3 min 12 s). Simulated iTBS will be administered using Magventure static cooling MCF-B65 coil.
  Arms: iTBS stimulation
Device: sham intermittent theta burst stimulation using a MagPro X100 — Patients randomized to receive sham iTBS will undergo the same procedure to patients receiving real iTBS. Sham iTBS will be administered using Magventure static cooling MCF-P-B65 coil that shares the same mechanical outline and produces identical sound level to MCF-B65 coil without stimulating the cerebral cortex.
  Arms: sham iTBS stimulation

SUMMARY:
Multiple sclerosis (MS) is a chronic and demyelinating disease of the central nervous system. It is one of the most common cause of neurological disability in young adults. Depression is a common symptom in MS patients, with lifetime prevalence rates going up to 50%. Depression not only reduces the response to treatment, delays the recovery of neurological function and social ability, but also significantly increases the risk of disability in patients with MS.

Transcranial magnetic stimulation (TMS) is a non-invasive method of brain stimulation that is based on electromagnetic induction. Intermittent theta burst stimulation (TBS), a newer form of rTMS, delivers 600 pulses in just 3 min, versus 37.5 min for conventional rTMS, but it has been shown to produce similar effects in patient with treatment-resistant depression.

To observe the effect and safety of iTBS on patients with MS and depression, we design a double-blind, randomized controlled study. Results of this research will inform on the efficiency of the TMS for the treatment of depression in MS patients, which will reduce the risk of disability and improve the quality of life.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic and demyelinating disease of the central nervous system. It is one of the most common cause of neurological disability in young adults. Depression is a common symptom in MS patients, with lifetime prevalence rates going up to 50%. Depression not only reduces the response to treatment, delays the recovery of neurological function and social ability, but also significantly increases the risk of disability in patients with MS. It is worth noting that depression remains widely underdiagnosed and untreated in MS patients. The investigators aim to treat the depression in MS patients using a non-invasive method, which will help improve life quality and reduce the risk of disability in patients.

Transcranial magnetic stimulation (TMS) is a non-invasive method of brain stimulation that uses magnetic fields to stimulate nerve cells in brain. Repetitive TMS (rTMS) is usually applied in antidepressant-resistant depression. Furthermore, some clinical trials show that rTMS also significantly improve Parkinson's related depression and postpartum depression. Intermittent theta burst stimulation (TBS), a newer form of rTMS, delivers 600 pulses in just 3 min, versus 37.5 min for conventional rTMS, but it has been shown to produce similar effects in patient with treatment-resistant depression.

In this study, thirty patients who meet the criteria will be included. They will then be randomly assigned into the SHAM or iTBS group for the study intervention. Patients and outcome assessors will be masked to treatment allocation. SHAM or iTBS will be delivered to stimulate left dorsalateral prefrontal cortex (DLPFC). The protocol includes 600 pulses per session: triplet 50 Hz bursts, repeated at 5 Hz; 2 s on and 8 s off. Each patient will receive 2 sessions per day over a period of 10 days (total of 20 sessions). After the treatment phase, patients will be followed up once after two weeks. The presence and severity of side effects will be assessed by the physician from the Department of Neurology. Before and after the iTBS or SHAM intervention and after two weeks of follow-up, primary and secondary measurements will be performed.

Results of this study will inform on the efficiency of the TMS for the treatment of depression in MS patients, which will reduce the risk of disability and improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 18 to 65
* 2) Male and female patients with clinically definite MS according to 2017 McDonald criteria
* 3) EDSS 0 to 6
* 4) Score between 11 and 30 on the Montgomery-Asberg Depression Rating Scale (MADRS) and stable antidepressants therapy > 1 months before enrollment and during the follow-up period
* 5) Informed consent of patients

Exclusion Criteria:

* 1) History of seizures (personal or family)
* 2) Comedication with neuroleptics or tricyclic antidepressants
* 3) bipolar disorder
* 4) Presence of other diseases of the nervous system (history of stroke, brain injury, brain tumor, increased intracranial pressure)
* 5) Significant neurologic, psychiatric, cardiovascular, hepatic, renal, gastrointestinal, metabolic, or other systemic comorbidities.
* 6) History of drug or alcohol abuse
* 7) Cardiac pacemakers
* 8) Metal implants in the head
* 9) Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) | 0 (baseline), 10 days and 4 weeks
  The MADRS is a 0-60 point scale to measure depression severity with a higher number indicating more severe depression. A score of 0-6 indicates symptoms absent, 7-19 indicates mild depression, 20-34 moderate, and > 34 severe.

SECONDARY OUTCOMES:
Presence and changes in severity of side effects | 0 (baseline), 10 days and 4 weeks
  Adverse events will be assessed by the physician from Department of Neurology weekly.
Change in Beck Depressive Inventory (BDI) | 0 (baseline), 10 days and 4 weeks
  BDI is a widely utilized to assess depression in MS patients. It is a 21-item self-reporting questionnaire for evaluating the severity of depression. The score range is 0-63 with higher scores indicating higher intensity.
Change in 21-item Beck's Anxiety Inventory (BAI) | 0 (baseline), 10 days and 4 weeks
  BAI is a self-report test for measuring anxiety severity and level. It contains 21 multiple-choice questions. The score range is 0-63 with higher scores indicating higher intensity.
Change in Fatigue Severity Scale (FSS) | 0 (baseline), 10 days and 4 weeks
  The FSS is a 9-item scale which measure the severity of fatigue and its effect on an individual's daily living and social participation. The total score ranges from 9 to 63, with a higher score indicate greater fatigue severity.
Change in Pittsburgh Sleep Quality Index (PSQI) | 0 (baseline), 10 days and 4 weeks
  PSQI is a self-rated questionnaire designed to evaluate overall sleep quality during the past month. Each of the questionnaire's 19 self-reported items belongs to one of seven subcategories: sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, use of sleep medication, degree of daytime dysfunction.
Change in Expand Disability Status Scale (EDSS) | 0 (baseline), 10 days and 4 weeks
  EDSS is a standardized method used to classify the severity and progression of multiple sclerosis. It provides a total score on a scale that ranges from 0 to 10.
Change in Cortical silent period (CSP) duration | 0 (baseline), 10 days and 4 weeks
  CSP duration will be measured by Magventure X100 + option.
Change in short-interval intracortical inhibition (SICI) | 0 (baseline), 10 days and 4 weeks
  SICI will be measured by Magventure X100 + option.
Change in intracortical facilitation (ICF) | 0 (baseline), 10 days and 4 weeks
  ICF will be measured by Magventure X100 + option.
Changes in long-interval intracortical inhibition (LICI) | 0 (baseline), 10 days and 4 weeks
  LICI will be measured by Magventure X100 + option.
Change in slow-wave/fast-wave (theta/beta) ratio from resting-state electroencephalograph (EEG) recording | 0 (baseline), 10 days and 4 weeks
  Resting-state EEG will be recorded by Nicolet EEG system.
Serum biomarker | 0 (baseline), 10 days
  Serum biomarker such as BDNF, TNF-alpha, IL-1 beta, S100 beta will be examined before and after TMS treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Qiu, MD/Ph.D, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University; Liqing Wang, MD/Ph.D, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoang H, Laursen B, Stenager EN, Stenager E. Psychiatric co-morbidity in multiple sclerosis: The risk of depression and anxiety before and after MS diagnosis. Mult Scler. 2016 Mar;22(3):347-53. doi: 10.1177/1352458515588973. Epub 2015 Jun 3. PMID 26041803
- [Background] Johansson V, Lundholm C, Hillert J, Masterman T, Lichtenstein P, Landen M, Hultman CM. Multiple sclerosis and psychiatric disorders: comorbidity and sibling risk in a nationwide Swedish cohort. Mult Scler. 2014 Dec;20(14):1881-91. doi: 10.1177/1352458514540970. Epub 2014 Jul 10. PMID 25013151
- [Background] Boeschoten RE, Braamse AMJ, Beekman ATF, Cuijpers P, van Oppen P, Dekker J, Uitdehaag BMJ. Prevalence of depression and anxiety in Multiple Sclerosis: A systematic review and meta-analysis. J Neurol Sci. 2017 Jan 15;372:331-341. doi: 10.1016/j.jns.2016.11.067. Epub 2016 Nov 30. PMID 28017241
- [Background] Siegert RJ, Abernethy DA. Depression in multiple sclerosis: a review. J Neurol Neurosurg Psychiatry. 2005 Apr;76(4):469-75. doi: 10.1136/jnnp.2004.054635. PMID 15774430
- [Background] Marrie RA, Fisk JD, Tremlett H, Wolfson C, Warren S, Tennakoon A, Leung S, Patten SB; CIHR Team in the Epidemiology and Impact of Comorbidity on Multiple Sclerosis. Differences in the burden of psychiatric comorbidity in MS vs the general population. Neurology. 2015 Dec 1;85(22):1972-9. doi: 10.1212/WNL.0000000000002174. Epub 2015 Oct 30. PMID 26519542
- [Background] Marrie RA, Walld R, Bolton JM, Sareen J, Patten SB, Singer A, Lix LM, Hitchon CA, El-Gabalawy R, Katz A, Fisk JD, Bernstein CN; CIHR Team in Defining the Burden and Managing the Effects of Psychiatric Comorbidity in Chronic Immunoinflammatory Disease. Psychiatric comorbidity increases mortality in immune-mediated inflammatory diseases. Gen Hosp Psychiatry. 2018 Jul-Aug;53:65-72. doi: 10.1016/j.genhosppsych.2018.06.001. Epub 2018 Jun 7. PMID 29929117
- [Background] McKay KA, Tremlett H, Fisk JD, Zhang T, Patten SB, Kastrukoff L, Campbell T, Marrie RA; CIHR Team in the Epidemiology and Impact of Comorbidity on Multiple Sclerosis. Psychiatric comorbidity is associated with disability progression in multiple sclerosis. Neurology. 2018 Apr 10;90(15):e1316-e1323. doi: 10.1212/WNL.0000000000005302. Epub 2018 Mar 9. PMID 29523642
- [Background] Binzer S, McKay KA, Brenner P, Hillert J, Manouchehrinia A. Disability worsening among persons with multiple sclerosis and depression: A Swedish cohort study. Neurology. 2019 Dec 10;93(24):e2216-e2223. doi: 10.1212/WNL.0000000000008617. Epub 2019 Nov 8. PMID 31704791
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Centonze D, Koch G, Versace V, Mori F, Rossi S, Brusa L, Grossi K, Torelli F, Prosperetti C, Cervellino A, Marfia GA, Stanzione P, Marciani MG, Boffa L, Bernardi G. Repetitive transcranial magnetic stimulation of the motor cortex ameliorates spasticity in multiple sclerosis. Neurology. 2007 Mar 27;68(13):1045-50. doi: 10.1212/01.wnl.0000257818.16952.62. PMID 17389310
- [Background] Gaede G, Tiede M, Lorenz I, Brandt AU, Pfueller C, Dorr J, Bellmann-Strobl J, Piper SK, Roth Y, Zangen A, Schippling S, Paul F. Safety and preliminary efficacy of deep transcranial magnetic stimulation in MS-related fatigue. Neurol Neuroimmunol Neuroinflamm. 2017 Dec 13;5(1):e423. doi: 10.1212/NXI.0000000000000423. eCollection 2018 Jan. PMID 29259998
- [Background] Hulst HE, Goldschmidt T, Nitsche MA, de Wit SJ, van den Heuvel OA, Barkhof F, Paulus W, van der Werf YD, Geurts JJG. rTMS affects working memory performance, brain activation and functional connectivity in patients with multiple sclerosis. J Neurol Neurosurg Psychiatry. 2017 May;88(5):386-394. doi: 10.1136/jnnp-2016-314224. Epub 2016 Dec 14. PMID 27974394